CLINICAL TRIAL: NCT05863663
Title: Examination of Chronic Pelvic Pain in Women With Endometriosis in the Context of the Degree of Physical Activity and Quality of Life
Brief Title: Chronic Pelvic Pain in Endometriosis
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 9534-PTE2023
Record Dates: First submitted 2023-04-12; First posted 2023-05-18 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Endometriosis; Physical Inactivity; Chronic Pelvic Pain Syndrome; Quality of Life
Keywords: endometriosis; pelvic pain; physical activity; chronic pain; health related quality of life
MeSH Terms: conditions — Endometriosis; Sedentary Behavior; Pelvic Pain; Motor Activity; Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endometriosis: Women diagnosed with endometriosis between 18-50 years old
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — cross sectional questionnaire

SUMMARY:
Endometriosis is a chronic, inflammatory disease affecting 10% (1 out of 10) of women of reproductive age. Pelvic pain is common among women with endometriosis.

Women with chronic pelvic pain conditions have elevated rates of relational stress and lower quality of life.

The aim of our study is to analyse the extent of pelvic pain associated with endometriosis, as well as the study focuses on correlations between pelvic pain and physical activity, pain-related self-efficacy, perceived stress and different aspects of health related quality of life.

DETAILED DESCRIPTION:
A cross-sectional study was conducted involving women with diagnosis of endometriosis.Patients with endometriosis and healthy women as controls are also recruited in the study.

The investigators used self-composed questionnaire for evaluating socio-demographic data and life-style factors, gynecological anamnesis, endometriosis diagnosis and further chronic conditions. Pain intensity was evaluated using Visual Analog Scale (VAS) focusing on perceived pain at present, the avarage perceived pain last month and the most intense perceived pain last month. Further measuring instruments were the Perceived Stress Scale (PSS) for evaluating stress levels among subjects, SF 36 short form health survey questionnaire for measuring health-related quality of life, Global Physical Activity Questionnaire (GPAQ) for evaluating physical activity of the subjects, Pain Catastrophizing Scale (PCS) for examining the subjects' perception of and reaction for a painful event, Pelvic Pain Impact Questionnaire (PPIQ) for evaluating the pelvic pain impact on the subjects' ability to perform physical activity, prolonged sitting, limitations in social activities, sexual activities and intimacy, Pain Self-Efficacy Questionnaire (PSEQ) for evaluating the confidence in performing different activities.

The participants are women between 18-50 years old and provided written informed consent. The investigators used convenience sampling method and the data were collected through online surveys. Data were analysed using IBM SPSS 28.0 and Microsoft Excel 2018 softwares and descriptive statistics, average, mean, standard deviation, two sample t-test, Pearson chi square test, Kolmogorov-Smirnov and Shapiro-Wilk test.

Dependent variables were the level of pelvic pain, physical activity, scores on the questionnairies, body mass index (BMI), independent variables were age, diagnosis of endometriosis, educational level.

In the course of this study, the cultural adaptation of the PSEQ questionnaire into Hungarian is also carried out based on Beaton's guidelines.

ELIGIBILITY:
Inclusion Criteria:

* women
* for study population: women diagnosed with endometriosis
* for control: women not diagnosed with endometriosis
* women between 18-50 years old
* signed informed consent

Exclusion Criteria:

* malignant tumor
* current pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between 18-50 years old and diagnosed with endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Pelvic pain | 1 day
  Visual Analogue Scale - 1-10 points; The more the points the severe the pain.
Pain self-efficacy | 1 day
  Pain self-efficacy questionnaire points Scale:0-60 Max points:60 Minimum points:0 The higher the point the better the condition is.
Physical activity | 1 day
  Global Physical Activity Questionnaire, min/week MET/week
Pelvic pain impact | 1 day
  Pelvic Pain Impact Questionnaire, Max points: 40 Minimum points: 0 Scale: higher points indicate higher impact on every day life
health-related quality of life | 1 day
  Short-Form 36 Questionnaire Subscales: physical functioning, role functioning/physical, role functioning/emotional, energy fatigue, emotional well-being, social functioning, pain, general health, health change
  Scoring is different between the items.
perceived stress | 1 day
  Perceived Stress Scale Scale: 0-40 Minimum points: 0 Maximum points:40 Scoring: Higher scores indicate high perceived stress Scores ranging from 0-13 are considered low perceived stress, ranging from 14-26 are considered moderate stress and ranging from 27-40 are considered high perceived stress

SECONDARY OUTCOMES:
Level of pain catastrophizing | 1 day
  Pain Catastrophizing Scale 13 questions ranging from 0-4 Minimum points: 0 Maximum points: 52 Higher points indicate higher level of pain catastrophizing
body mass index | 1 day
  BMI kg/m2
level of education | 1 day
  what is your educational level? 4 types of answer
  * unfinished elementary school
  * finished elementary school
  * high school
  * bachelor/masters degree
Endometriosis and menstrual pain | 1 day
  Endopain 4D Questionnaire
  The ENDOPAIN-4D comprises 21 items divided into four subparts: spontaneous pelvic pain and dysmenorrhoea (questions 1 to 10), dyspareunia (questions 11 to 13), intestinal pain symptoms (questions 14 to 16), and other symptoms (questions 17 to 21). Each question is first scored dichotomously as yes/no.
lifestyle factors | 1 day
  Questions about alcohol intake, smoking, nutritional habits
  Open ended questions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kovacs-Szabo Z, Acs P, Makai A, Hock M. Validity and reliability testing of the Pelvic Pain Impact Questionnaire. Sci Rep. 2025 Oct 3;15(1):34628. doi: 10.1038/s41598-025-18269-3. PMID 41044332